CLINICAL TRIAL: NCT00726739
Title: A Randomized Phase II Study of IL-2 With or Without an Allogeneic Large Multivalent Immunogen (LMI) Vaccine for the Treatment of Stage IV Melanoma
Brief Title: Aldesleukin With or Without Vaccine Therapy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2006LS046; UMN-0701M01001 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-07-31; First posted 2008-08-01 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Stage IV Melanoma
Keywords: recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I - LMI + aldesleukin (Experimental): Patients receive allogeneic large multivalent immunogen vaccine (LMI) LP2307 intradermally on day 1 and aldesleukin subcutaneously (SC) on days 7 and 8. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: aldesleukin; Biological: allogeneic large multivalent immunogen vaccine
- Arm II (control) - aldesleukin (Active Comparator): Patients receive aldesleukin SC on days 1 and 2. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross over and receive treatment on arm I.
  Interventions: Biological: aldesleukin
- Arm III - Crossover Patients (Experimental): Patients who have progressive disease on Arm II were be offered crossover to Arm I provided they continued to meet all study criteria.
  Patients receive allogeneic large multivalent immunogen vaccine (LMI) LP2307 intradermally on day 1 and aldesleukin subcutaneously (SC) on days 7 and 8. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Biological: aldesleukin; Biological: allogeneic large multivalent immunogen vaccine

INTERVENTIONS:
Biological: aldesleukin — IL-2 Alone - administer 10 x 10^6 International Units subcutaneously (SQ) will be given on day 1 and day 2 every 4 weeks until disease progression or for a maximum of 12 treatment cycles.
  Other Names: IL-2; Interleukin-2; Proleukin
Biological: allogeneic large multivalent immunogen vaccine — Allogeneic tumor cell membrane-coated large multivalent immunogen (LMI [1 x 10^7, 5-μm silica spheres]) will be given as an intradermal injection every 4 weeks for up to 12 injections. Each vaccine dose will be 0.2 ml.
  Other Names: LMI vaccine
  Arms: Arm I - LMI + aldesleukin; Arm III - Crossover Patients

SUMMARY:
RATIONALE: Aldesleukin may stimulate the white blood cells to kill tumor cells. Vaccines may help the body build an effective immune response to kill tumor cells. Giving aldesleukin together with vaccine therapy may kill more tumor cells. It is not yet known whether aldesleukin is more effective with or without vaccine therapy in treating melanoma.

PURPOSE: This randomized phase II trial is studying how well aldesleukin works when given with or without vaccine therapy in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the progression-free survival of patients with stage IV melanoma treated with aldesleukin with vs without allogeneic large multivalent immunogen melanoma vaccine LP2307.

Secondary

* To compare the clinical response in patients treated with these regimens.
* To compare the 1- and 2-year survival rates in patients treated with these regimens.
* To determine whether an immune response is generated after vaccination in these patients.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive allogeneic large multivalent immunogen melanoma vaccine LP2307 intradermally on day 1 and aldesleukin subcutaneously (SC) on days 7 and 8. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (control): Patients receive aldesleukin SC on days 1 and 2. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross over and receive treatment on arm I.

Patients undergo blood sample collection periodically for correlative laboratory studies. Samples are analyzed for immune responses to keyhole limpet hemocyanin and tetanus toxoid (control antigens) by ELISA assay; IFN-γ production by CD8 T cells in response to melanoma-derived peptides by ELISpot assay; delayed-type hypersensitivity response to vaccination; and frequency of peripheral blood lymphocytes, including T cells, B cells, NK cells, and monocytes, by flow cytometry.

* Arm III Crossover: Patients who have progressive disease on Arm II will be offered crossover to Arm I provided they continue to meet all study criteria.

After completion of study treatment, patients are followed every 2 months for 1 year, every 3 months until disease progression, and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV melanoma.
* Prior systemic chemotherapy, immunotherapy, or biological therapy is allowed if at least 4 weeks since last treatment. Patient must recover from the acute toxic effects of the treatment prior to study enrollment.
* Disease status must be that of measurable or nonmeasurable disease as defined by Solid Tumor Response Criteria (RECIST)
* Karnofsky performance status >70% (Eastern Cooperative Oncology Group 0-1)
* Age 18 years or older
* Adequate organ function within 14 days of study enrollment including the following:

  * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 10^9/L, platelets ≥100 x 10^9/L, and hemoglobin ≥ 10 g/dL
  * Hepatic: bilirubin < 3 times the upper limit of normal (× ULN), aspartate transaminase (AST) < 3 × ULN
  * Renal: creatinine ≤ 2.0
* Must share at least one class I HLA allele with the HLA-type SK23-CD80+ cell (class I alleles (A1, A2, B7, B8, C7))
* Meets eligibility criteria for and agrees to enroll in "MT1999- 06: Vaccination with Tetanus Toxoid and Keyhole Limpet Hemocyanin (KLH) to Assess Antigen-Specific Immune Responses" (IRB # 9904M01581, CPRC #2002LS032)
* Women of childbearing potential and men whose partners are of childbearing potential are required to use an effective method of contraception (ie, a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study and for 3 months after the last dose of study drug.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion criteria:

* History of brain metastases or positive brain scan at on-study
* Immunosuppressive therapy i.e., prednisone or organ transplant patients, however topical or inhalational steroids are allowed.
* Autoimmune diseases requiring immunosuppressive therapy.
* History of symptomatic pulmonary disease will have pulmonary function tests (PFTs) performed. Patients with symptoms of dyspnea or rales, wheezes or rhonchi on physical exam will undergo PFTs. Those with FEV1 <50% of predicted or corrected DLCO <50% are not eligible.
* Patients with cardiac disease such as recent myocardial infarction (< 3 months prior), unstable angina, or heart failure requiring medical intervention will undergo cardiac evaluation. Cardiac testing may include ECG, MUGA or echocardiogram, and/or thallium stress test as indicated to evaluate cardiac risks. Those patients with exercise-induced ischemia or an ejection fraction by MUGA or echocardiogram < 40% are not eligible.
* Due to the origin of the KLH protein, patients with a history of seafood allergy are excluded from receiving KLH.
* Hypersensitivity to any component of the vaccine, including Thimerosal, a mercury derivative, is a contraindication (taken from tetanus toxoid package insert).
* The occurrence of any type of neurologic symptoms to tetanus vaccine in the past is a contraindication to further use (taken from tetanus toxoid package insert).
* Subjects who have had tetanus toxoid within the last 7 years will not receive the tetanus vaccine component of this
* Pregnant (positive pregnancy test) or lactating women. Use of LMI vaccine during pregnancy is not approved for use by the FDA during pregnancy. IL-2 is pregnancy category C - risk in pregnancy cannot be ruled out.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were evaluated for eligibility by one of the investigators prior to enrollment.
Pre-assignment Details: This study requires concurrent registration to the University of Minnesota study "MT1999-06: Vaccination with Tetanus Toxoid and Keyhole Limpet Hemocyanin (KLH) to Assess Antigen-Specific Immune Responses" (IRB # 9904M01581, CPRC #2002LS032).
Groups:
- Arm I and III Crossover Group - LMI + Aldesleukin: Patients receive allogeneic large multivalent immunogen melanoma vaccine (LMI) LP2307 intradermally on day 1 and aldesleukin subcutaneously (SC) on days 7 and 8. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Includes 6 patients who progressed and "crossed over" from Arm II.
Period: Overall Study
Arm/Group | Arm I and III Crossover Group - LMI + Aldesleukin | Arm II (Control) - Aldesleukin
Started | 11 | 10
Completed | 10 (1 patient failed during screening due to brain metastasis.) | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I and III Crossover Group - LMI + Aldesleukin: Includes 6 patients who progressed and "crossed over" from Arm II.
- Total: Total of all reporting groups
Arm/Group | Arm I and III Crossover Group - LMI + Aldesleukin | Arm II (Control) - Aldesleukin | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.4) | 64.0 (14.9) | 63.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Median Time of Progression-free Survival
Description: Progression free survival (PFS) was measured in months from date of randomization to date of disease progression, or date of death. For patients who died without tumor progression, PFS assumes their deaths are randomly related to tumor progression. Therefore, PFS includes deaths if they came first.
Time Frame: From Date of Randomization to Date of Disease Progression or Last Contact - up to 2 years.
Population: All patients who received at least one dose of study treatment are included. One patient who was originally screened and randomized did not receive treatment due to brain metastasis. This patient was included in PFS analysis based on the intent-to-treat principle, but was excluded from the evaluation of adverse events.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm I and III Crossover Group - LMI + Aldesleukin | Arm II (Control) - Aldesleukin
Number analyzed (Participants) | 11 | 10
Months | 2.20 [0.03 to 4.07] | 1.95 [0.95 to 20.60]

2. Secondary Outcome: Clinical Response of Lesion(s)
Description: Beginning at 2 months Through End of Treatment: To determine clinical response of each treatment group - Best Clinical response will be determined using Solid Tumor Response Criteria (RECIST). Complete Response (CR) = complete disappearance of all target lesions. Partial Response (PR) = At least a 30% decrease in sum of longest diameters of target lesions. Progressive Disease (PD) = At least a 20% increase in sum of longest diameters of target lesions. Stable Disease (SD) = Neither sufficient shrinkage to qualify for PR or PD.
Time Frame: Month 2 through Month 12
Population: All patients who received at least one dose of study treatment are included. One patient who was originally screened did not receive treatment due to brain metastasis.
Measure: Number; unit: participants
Arm/Group | Arm I and III Crossover Group - LMI + Aldesleukin | Arm II (Control) - Aldesleukin
Number analyzed (Participants) | 11 | 10
participants
  Complete Response (CR) | 0 | 1
  Partial Response (PR) | 0 | 0
  Stable Disease (SD) | 2 | 1
  Progressive Disease (PD) | 8 | 8
  Missing information | 1 | 0

3. Secondary Outcome: Overall Survival at 2 Years
Description: Two year survival (alive at 2 years from randomization) rate of each treatment group.
Time Frame: 2 Years
Measure: Number; unit: percentage of patients
Arm/Group | Arm I and III Crossover Group - LMI + Aldesleukin | Arm II (Control) - Aldesleukin
Number analyzed (Participants) | 11 | 10
percentage of patients | 24 | 27

4. Secondary Outcome: Overall Survival at 1 Year
Description: One year survival (alive at 1 year from randomization) rate of each treatment group.
Time Frame: 1 Year
Measure: Number; unit: Percentage of patients
Arm/Group | Arm I and III Crossover Group - LMI + Aldesleukin | Arm II (Control) - Aldesleukin
Number analyzed (Participants) | 11 | 10
Percentage of patients | 45 | 40

5. Secondary Outcome: Immune Response
Description: Immune responses is be assessed by Delayed Type Hypersensitive (DTH) responses to LMI, IFN-γ production by CD8 T cells using the ELISPOT assay, and CD8 T cell binding to HLA-A2 multimers complexed with melanoma-derived peptides (pentamer analysis). DTH reactions are determined at 48 hours by measuring the largest diameter and right angle diameter of the area of induration and calculating the mean. DTH responses are recorded as present or absent but cannot be used as a quantitative measure of immune activation.
Time Frame: 48 hours After Study Medication
Measure: Number; unit: participants
Groups:
- Arm I and III Crossover Group - LMI + Aldesleukin: Patients receive allogeneic large multivalent immunogen melanoma vaccine (LMI) LP2307 intradermally on day 1 and aldesleukin subcutaneously (SC) on days 7 and 8. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Includes 6 patients who progressed and "crossed over" from Arm II. Both KLH and DTH are tests assessing the ability to respond to immune therapy. These are independent tests and there is no bearing of KLH response on DTH response.
Arm/Group | Arm I and III Crossover Group - LMI + Aldesleukin | Arm II (Control) - Aldesleukin
Number analyzed (Participants) | 11 | 10
participants
  KLH twofold responder | 5 | 8
  KLH tenfold responder | 2 | 7
  Missing information | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 28 days (+/- 14 day) after last dose of study drug, an average of 1 year.
Description: One patient withdrew after randomization and before LMI (large multivalent immunogen) +IL2 (aldesleukin) started and was excluded from the evaluation of toxicity (Arm I group).
Arm/Group | Arm I and III Crossover Group - LMI + Aldesleukin | Arm II (Control) - Aldesleukin
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/10
Other Adverse Events (participants affected / at risk) | 4/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I and III Crossover Group - LMI + Aldesleukin (N=10) | Arm II (Control) - Aldesleukin (N=10)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Supraventricular and nodal arrhythmia
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain - back (General disorders) | 1 (1) | 0 (0)
Progressive Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I and III Crossover Group - LMI + Aldesleukin (N=10) | Arm II (Control) - Aldesleukin (N=10)
Allergic reaction, hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood/bone marrow, other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatology/skin, other (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (heartburn) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (10)
Dyspnea, shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Edema, peripheral (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fever (in absence of neutropenia) (Infections and infestations) | 1 (1) | 0 (0)
Flu-like syndrome (General disorders) | 0 (0) | 2 (2)
Gastrointestinal, other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hemorrhage, respiratory tract (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection with normal ANC, Urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC, blood (Infections and infestations) | 1 (1) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)
Mucositis (oral cavity (Gastrointestinal disorders) | 1 (1) | 1 (1)
Muscle weakness, generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (3)
Neuropathy, cranial (Nervous system disorders) | 0 (0) | 1 (1) — CN IX motor-pharynx, sensory-ear, pharynx, tongue
Pain, abdomen (General disorders) | 2 (2) | 1 (1)
Pain, chest wall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain, headache (General disorders) | 0 (0) | 1 (1)
Pain, other (General disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pulmonary respiratory, other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rash, desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Voice changes, hoarseness (Gastrointestinal disorders) | 0 (0) | 1 (1) — laryngitis
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes